CLINICAL TRIAL: NCT01676779
Title: Randomized Controlled Phase II Clinical Trial on mRNA Electroporated Autologous Dendritic Cells for Stage III/IV Melanoma Patients Who Are Disease-free Following the Local Treatment of Macrometastases.
Brief Title: mRNA Electroporated Autologous Dendritic Cells for Stage III/IV Melanoma
Acronym: DC-MEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: RIZIV (Unknown)
Responsible Party: Principal Investigator, Bart Neyns, Head of devision (Medical Oncology), Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC-MEL
Record Dates: First submitted 2012-08-21; First posted 2012-08-31 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Malignant Melanoma Stage III; Malignant Melanoma Stage IV
Keywords: melanoma; no evidence of disease; resection; macro-metastases
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A dendritic cell therapy (Experimental): Arm-A, patients will receive Dendritic Cell therapy during one year following randomization.
  Interventions: Biological: Dendritic cell therapy
- Arm B Dendritic cell therapy (Experimental): Arm-B, patients will initiate Dendritic Cell therapy only after documented recurrence of the melanoma that cannot be salvaged by local therapy.
  Interventions: Biological: Dendritic cell therapy

INTERVENTIONS:
Biological: Dendritic cell therapy — Dendritic cell therapy IV and ID

SUMMARY:
This is an open label, 2-arm, 1-stage, randomized controlled phase II study in patients with AJCC stage IIIB/C & -IV melanoma. At baseline tumor assessment (using total body FDG-PET/CT), patients should be free from measurable tumor lesions (according to RECISTv1.1 definitions) following prior local therapy (e.g. following surgical resection, isolated limb perfusion, radiofrequency ablation, cryotherapy, radiotherapy, electrochemotherapy, …). Patients should not have symptomatic non-measurable tumor lesions (e.g. bone metastasis, or pleural effusion), and lesions treated by prior local therapy should be free from progression. Patients should not have received any prior systemic therapy (non-experimental or experimental).

DETAILED DESCRIPTION:
This is an open label, 2-arm, 1-stage, randomized controlled phase II study in patients with AJCC stage IIIB/C & -IV melanoma. At baseline tumor assessment (using total body FDG-PET/CT), patients should be free from measurable tumor lesions (according to RECISTv1.1 definitions) following prior local therapy (e.g. following surgical resection, isolated limb perfusion, radiofrequency ablation, cryotherapy, radiotherapy, electrochemotherapy, …). Patients should not have symptomatic non-measurable tumor lesions (e.g. bone metastasis, or pleural effusion), and lesions treated by prior local therapy should be free from progression. Patients should not have received any prior systemic therapy (non-experimental or experimental).

* Patients will be randomized between two treatment arms (Arm-A and -B). In study Arm-A, patients will receive DC-administrations during one year following randomization. Salvage treatment by local therapies will be allowed during the study treatment in Arm-A. In study Arm-B, patients will initiate DC-administrations only after documented recurrence of the melanoma that cannot be salvaged by local therapy.
* The primary endpoint of this clinical trial is to determine the rate (%) of patients who are free from macrometastases (: measurable tumor lesions and symptomatic non-measurable tumor lesions) at 1-year (= 52 weeks) after randomization.

Patients treated on Arm-B will serve as a contemporary control-arm to help interpreting the outcome of patients treated in Arm-A. By design (phase II) this trial will not be powered to statistically prove a predefined difference between the two study arms (this would require a phase III design). Patients treated in Arm-B will be able to initiate immunotherapy with autologous DC at the time of recurrence that can not be salvaged by local therapy. Documentation of the anti-tumor activity and survival following DC-treatment at recurrence in Arm-B patients will be a secondary objective of this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent
2. Histological documentation of AJCC stage III or stage IV melanoma
3. melanoma (melanoma originating in the choroid, iris or ciliar body are not eligible)
4. baseline tumor assessment by whole-body FDG-PET/CT, patients should be free from measurable tumor lesions (RECIST (v1.1)), and free from symptomatic non-measurable tumor lesions
5. Prior local treatment of primary and metastatic tumor lesions is allowed . Treated tumor lesions should be free from progression at baseline assessment
6. Normal organ function and normal hematological parameters;laboratory parameters should be within normal range, except following laboratory parameters:HEMOGLOBIN ≥ 10 G/DL; GRANULOCYTES ≥ 1,500/µL; LYMPHOCYTES ≥ 1000/µL; PLATELETS ≥ 100,000/µL; SERUM CREATININ ≤ 2.0 MG/DL; SERUM BILIRUBIN ≤ 2.0 MG/DL; AST AND ALT ≤ 2 X THE NORMAL UPPER LIMITS; LDH ≤ 1,5X NORMAL UPPER LIMIT; CRP ≤ 1,5X NORMAL UPPER LIMIT; PROTHROMBIN TIME (PT) INTERNATIONAL NORMALIZED RATIO (INR) AND PARTIAL THROMBOPLASTIN TIME (PTT) WITHIN NORMAL LIMITS
7. Negative serology for HCV, and HIV; absence of active infection with HBV, and Syphilis; If positive results for HepB or Syphilis indicate immunity and are not indicative of active infection, the patient can enter the study.
8. Adequate venous access(to undergo leukapheresis)
9. No prior systemic therapy for melanoma
10. Full recovery from all prior therapies. A period of 4 weeks following major surgery, radiation therapy, or ILP, or any other major invasive procedure is required
11. Baseline WHO performance status of 0 or 1
12. Male and female patients ≥ 18 years
13. No need for uninterrupted therapeutic anticoagulation
14. No prior history of a serious autoimmune disorder
15. No concomitant medication with immune suppressive drugs
16. Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

1. Evidence of immunodeficiency or autoimmune disease requiring medical treatment (e.g. corticosteroids or other immunosuppressive drugs).Vitiligo is not an exclusion criterion
2. Any serious acute or chronic illnesses (e.g. heart disease NYHA Class III or IV,renal-,liver- or pulmonary insufficiency) or other conditions requiring concurrent medications not allowed during this study (e.g. active chronic infections requiring antibiotics)
3. History of malignancy. Curatively treated cervical carcinoma in situ,or squamous-,or basal cell carcinoma of the skin, or subjects who have been treated and recurrence-free of other malignancies for more than 5 years following the diagnosis are eligible
4. Inability to undergo FDG-PET/CT, or MRI examination
5. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
6. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment
7. Subject is pregnant (positive serum beta-HCG test at screening) or is currently breast-feeding, anticipates becoming pregnant/impregnating their partner during the study or within 6 months after study participation, or subject does not agree to follow acceptable methods of birth control, to avoid conception during the study and for at least 6 months after receiving the last dose of study treatment
8. Current alcohol dependence or drug abuse
9. Known hypersensitivity to the study treatment
10. Legal incapacity or limited legal capacity
11. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
12. Signs and symptoms suggestive of transmissible spongiform encephalopathy,or family members who suffer(ed) from such.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
1-year disease free survival percentage | 1-year following recruitment date
  Patients will be evaluated 52 weeks following randomization for their melanoma disease status (= macro-metastases present or absent)

SECONDARY OUTCOMES:
safety | continuous during the study (52weeks after start)
  Patients will be followed continuous during their study participation for adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, Phd Md, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium